CLINICAL TRIAL: NCT02728206
Title: A Phase 2, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir/Velpatasvir Fixed Dose Combination Administered for Four Weeks in Patients Infected With Chronic HCV in the Peri-Operative Liver Transplantation Setting
Brief Title: Sofosbuvir/Velpatasvir Fixed-Dose Combination in HCV-Infected Adults Who Are Undergoing Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-2083
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SOF/VEL (Experimental): SOF/VEL FDC for 4 weeks starting on the day of or day after the participant's liver transplant
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) in hepatitis C virus (HCV)-infected adults who are undergoing liver transplantation.

ELIGIBILITY:
Key Inclusion Criteria:

* HCV-infected, male and non-pregnant/non-lactating females, who are undergoing liver transplantation

Key Exclusion Criteria:

* Receiving an HCV-infected liver
* HIV or hepatitis B virus (HBV) co-infected

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-12 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a study site in New Zealand. The first participant was screened on 12 June 2016. The last study visit occurred on 16 January 2018.
Pre-assignment Details: 11 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily for 4 weeks starting on the day of or day after the participant's liver transplant.
Period: Overall Study
Arm/Group | SOF/VEL
Started | 9
Completed | 8
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet orally once daily for 4 weeks starting on the day of or day after the participant's liver transplant.
Arm/Group | SOF/VEL
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Pre-Transplant Hepatitis C Virus (HCV) genotype [Count of Participants; unit: Participants]
  Genotype 1a | 2
  Genotype 1/1b | 1
  Genotype 3 | 5
  Genotype 3a | 1
Pre-Transplant IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 8
    CT | 1
Pre-Transplant HCV RNA (log10 international units per milliliter (IU/mL)) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.4 (0.63)
Pre-Transplant HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 3
  ≥ 800,000 IU/mL | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all enrolled participants who received a liver transplant, and took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 9
Percentage of participants | 77.8 [40.0 to 97.2]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to Week 4
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 9
Percentage of participants | 11.1

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 9
Percentage of participants | 88.9 [51.8 to 99.7]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment
Time Frame: Days 3, 5, 7, 14, 21, and 28
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 9
Percentage of participants
  Day 3 | 0 [0.0 to 33.6]
  Day 5 | 0 [0.0 to 33.6]
  Day 7 | 0 [0.0 to 33.6]
  Day 14 | 33.3 [7.5 to 70.1]
  Day 21: number analyzed (Participants) | 7
  Day 21 | 85.7 [42.1 to 99.6]
  Day 28: number analyzed (Participants) | 7
  Day 28 | 85.7 [42.1 to 99.6]

5. Secondary Outcome: Percentage of Participants With Overall Virologic Failure
Description: Virologic failure was defined as 1) End of Treatment Virologic Failure: HCV RNA ≥ 15 IU/mL at last observed HCV RNA measurement on or prior to last dose date of SOF/VEL + 3 days after completion of 28 ± 3 days of SOF/VEL treatment, or 2) Relapse: HCV RNA ≥ 15 IU/mL during the posttreatment follow-up period having achieved HCV RNA < 15 IU/mL at the end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement.
Time Frame: Up to Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 9
Percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks plus 30 days
Description: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | SOF/VEL
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=9)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Liver transplant rejection (Immune system disorders) | 3
Cytomegalovirus infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 2
Fluid intake reduced (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intensive care unit acquired weakness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=9)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Vision blurred (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oedema (General disorders) | 1
Liver transplant rejection (Immune system disorders) | 3
Herpes simplex (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Bacterial test positive (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT02728206/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02728206/SAP_001.pdf